CLINICAL TRIAL: NCT05823493
Title: Schroth Exercises Combined With Laser Acupuncture Therapy
Brief Title: Effect of Schroth Exercises Combined With Laser Acupuncture Therapy in Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalian Second People's Hospital (Other)
Responsible Party: Principal Investigator, Guangyu Fu, Doctor, Dalian Second People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DLSP001
Record Dates: First submitted 2023-03-19; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Adolescent Idiopathic Scoliosis; Laser Acupuncture
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experimental group (Experimental)
  Interventions: Behavioral: Schroth exercise therapy; Device: laser therapy
- the control group (Active Comparator)
  Interventions: Behavioral: Schroth exercise therapy

INTERVENTIONS:
Behavioral: Schroth exercise therapy — The Schroth classification criteria includes four curve patterns that are determined with reference to the location of the curves, the importance of lumbar and thoracic prominences, and the effect of the scoliosis on the pelvis.
Device: laser therapy — Laser therapy was performed w ith a dual wavelength, high power IR laser (Multiwave Locked System (MLS®) laser, Mphi, ASA srl, Vicenza, Italy) and the laser acupuncture points include DU2, GB30, DU9, SP6, LR8, DU6, DU4, DU12. Laser puncture acupuncture points had been identified according to Traditional Chinese Medicine (TCM) and treated with handpiece optical group following the detailed treatment parameters: 900Hz, FPW mode, 60 s per point, 29.12J, spot size 3 cm2, energy density 27J/cm2. All treatments are performed five times in a week for 4 consecutive weeks.
  Arms: the experimental group

SUMMARY:
The goal of this clinical trial] is to explore the clinical effect of laser acupuncture combined with Schroth training on adolescent idiopathic scoliosis (AIS) . The main question[s] it aims to answer are:

* The effects of Schroth exercises on Cobb angles, angle of trunk rotation, spinal mobility, gait parameters and clinical efficacy in patients with AIS.
* Laser acupuncture combined with Schroth method on Cobb angles, angle of trunk rotation, spinal mobility, gait parameters and clinical efficacy in patients with AIS.

Participants will received Schroth exercise therapy and laser acupuncture therapy (MLS laser).

If there is a comparison group: Researchers will compare received Schroth exercise therapy to see the effects of Schroth exercises and laser acupuncture combined with Schroth method on Cobb angles, angle of trunk rotation, spinal mobility, gait parameters and clinical efficacy in patients with AIS

DETAILED DESCRIPTION:
In this study, the standard control, control group receipts schroth exercise therapy, while trial group receives Schroth exercise therapy and laser therapy. The design of the individual Schroth exercise is carried out according to the c urve patterns of the Schroth classification. The Schroth classification criteria includes four curve patterns that are determined with reference to the location of the curves, the importance of lumbar and thoracic prominences, and the effect of the scoliosis on the pelvis. Laser therapy was performed w ith a dual wavelength, high power IR laser (Multiwave Locked System (MLS®) laser, Mphi, ASA srl, Vicenza, Italy) and the laser acupuncture points include DU2, GB30, DU9, SP6, LR8, DU6, DU4, DU12. Laser puncture acupuncture points had been identified according to Traditional Chinese Medicine (TCM) and treated with handpiece optical group following the detailed treatment parameters: 900Hz, FPW mode, 60 s per point, 29.12J, spot size 3 cm2, energy density 27J/cm2. All treatments are performed five times in a week for 4 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent idiopathic scoliosis patients without history of traumas
* positive Adam's Forward Bend Test, Cobb Angle>10°

Exclusion Criteria:

* functional scoliosis and other structural scoliosis
* Previous history of scoliosis surgery
* Wearing braces and being treated in other ways
* Unable to complete PSSE training actions as required
* Complicated with serious heart, liver, kidney and other systemic diseases

Ages: 125 Months to 200 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Cobb angle(°) | before the whole treatment cycle
  Draw a line through the spine on the upper surface of the upper vertebra and the lower surface of the lower vertebra on the X-ray film, and make the vertical line of the above two lines, and measure the angle between the two vertical lines. All radiographs are measured three times by a professional physician with the same protractor, and the average value is recorded
Cobb angle(°) | 6 months after treatment
  Draw a line through the spine on the upper surface of the upper vertebra and the lower surface of the lower vertebra on the X-ray film, and make the vertical line of the above two lines, and measure the angle between the two vertical lines. All radiographs are measured three times by a professional physician with the same protractor, and the average value is recorded
Cobb angle(°) | 12 months after treatment
  Draw a line through the spine on the upper surface of the upper vertebra and the lower surface of the lower vertebra on the X-ray film, and make the vertical line of the above two lines, and measure the angle between the two vertical lines. All radiographs are measured three times by a professional physician with the same protractor, and the average value is recorded
Trunk rotation angle(°) | before the whole treatment cycle
  Trunk rotation angle (ATR) is measured with scoliosis instrument to quantitatively evaluate the chest rotation angle and waist rotation angle.
Trunk rotation angle(°) | 6 months after treatment
  Trunk rotation angle (ATR) is measured with scoliosis instrument to quantitatively evaluate the chest rotation angle and waist rotation angle.
Trunk rotation angle(°) | 12 months after treatment
  Trunk rotation angle (ATR) is measured with scoliosis instrument to quantitatively evaluate the chest rotation angle and waist rotation angle.
Musculoskeletal stiffness | before the whole treatment cycle
  Use PulStarG3 system (Sense Technology Inc) to evaluate the musculoskeletal stiffness of each spinal segment. The handheld pulse head presses on the patient and provides a single low-energy pulse to the vertebral layer of interest. The force sensor in the pulse head measures the resistance to the pulse and transmits the analysis results to a digital computer, which can be considered as a computer-assisted spinal palpation in a series of bar graphs (abnormal musculoskeletal hardness is shown in the red bar and normal musculoskeletal hardness is shown in the green bar).
Musculoskeletal stiffness | 6 months after treatment
  Use PulStarG3 system (Sense Technology Inc) to evaluate the musculoskeletal stiffness of each spinal segment. The handheld pulse head presses on the patient and provides a single low-energy pulse to the vertebral layer of interest. The force sensor in the pulse head measures the resistance to the pulse and transmits the analysis results to a digital computer, which can be considered as a computer-assisted spinal palpation in a series of bar graphs (abnormal musculoskeletal hardness is shown in the red bar and normal musculoskeletal hardness is shown in the green bar).
Musculoskeletal stiffness | 12 months after treatment
  Use PulStarG3 system (Sense Technology Inc) to evaluate the musculoskeletal stiffness of each spinal segment. The handheld pulse head presses on the patient and provides a single low-energy pulse to the vertebral layer of interest. The force sensor in the pulse head measures the resistance to the pulse and transmits the analysis results to a digital computer, which can be considered as a computer-assisted spinal palpation in a series of bar graphs (abnormal musculoskeletal hardness is shown in the red bar and normal musculoskeletal hardness is shown in the green bar).
Gait(stride length (m)) | before the whole treatment cycle
  collected by wearable devices (micro-electro-mechanical systems, MEMS), the sampling frequency is set at 20 Hz, and transmitted to the computer server according to the manufacturer's protocol. The collected gait parameters include average pressure distribution, stride length, stride length and walking speed.
Gait(stride time(s)) | before the whole treatment cycle
  collected by wearable devices (micro-electro-mechanical systems, MEMS), the sampling frequency is set at 20 Hz, and transmitted to the computer server according to the manufacturer's protocol. The collected gait parameters include average pressure distribution, stride length, stride length and walking speed.
Gait(walking speed(m/s)) | before the whole treatment cycle
  collected by wearable devices (micro-electro-mechanical systems, MEMS), the sampling frequency is set at 20 Hz, and transmitted to the computer server according to the manufacturer's protocol. The collected gait parameters include average pressure distribution, stride length, stride length and walking speed.
Gait(stride length (m)) | 6 months after treatment
  collected by wearable devices (micro-electro-mechanical systems, MEMS), the sampling frequency is set at 20 Hz, and transmitted to the computer server according to the manufacturer's protocol. The collected gait parameters include average pressure distribution, stride length, stride length and walking speed.
Gait(stride time(s)) | 6 months after treatment
  collected by wearable devices (micro-electro-mechanical systems, MEMS), the sampling frequency is set at 20 Hz, and transmitted to the computer server according to the manufacturer's protocol. The collected gait parameters include average pressure distribution, stride length, stride length and walking speed.
Gait(walking speed(m/s)) | 6 months after treatment
  collected by wearable devices (micro-electro-mechanical systems, MEMS), the sampling frequency is set at 20 Hz, and transmitted to the computer server according to the manufacturer's protocol. The collected gait parameters include average pressure distribution, stride length, stride length and walking speed.
Gait(stride length (m)) | 12 months after treatment
  collected by wearable devices (micro-electro-mechanical systems, MEMS), the sampling frequency is set at 20 Hz, and transmitted to the computer server according to the manufacturer's protocol. The collected gait parameters include average pressure distribution, stride length, stride length and walking speed.
Gait(stride time(s)) | 12 months after treatment
  collected by wearable devices (micro-electro-mechanical systems, MEMS), the sampling frequency is set at 20 Hz, and transmitted to the computer server according to the manufacturer's protocol. The collected gait parameters include average pressure distribution, stride length, stride length and walking speed.
Gait(walking speed(m/s)) | 12 months after treatment
  collected by wearable devices (micro-electro-mechanical systems, MEMS), the sampling frequency is set at 20 Hz, and transmitted to the computer server according to the manufacturer's protocol. The collected gait parameters include average pressure distribution, stride length, stride length and walking speed.

CONTACTS AND LOCATIONS:
Locations (1):
- Dalian Second People's Hospital, Dalian, China

IPD SHARING:
Plan to Share IPD: No